CLINICAL TRIAL: NCT03916276
Title: Mechanisms of Psychosocial Treatments on Opioid Use in Chronic Pain
Brief Title: Living in Full Even With Pain Study
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); The University of Queensland (Other); Medical University of South Carolina (Other); Rush University (Other)
Responsible Party: Principal Investigator, Mark Jensen, Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006474; R01AT008559-02S1 (NIH)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: Chronic Pain; Opioid; Heterogeneous Pain; Musculoskeletal Pain; Mindfulness Meditation; Behavioral Activation; Cognitive Therapy; Telehealth; Opioid Misuse; Mechanisms
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Opioid-Related Disorders | interventions — Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized 3-group, 90-subject clinical trial to test the mediators and moderators of cognitive therapy, mindfulness meditation, and behavioral activation on individuals with heterogeneous chronic pain conditions who are at risk for opioid misuse.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Therapy (CT) Condition (Active Comparator): Participants randomized to this arm will be taught to recognize the relationships between thoughts, feelings, behaviors, and pain. This technique will help participants: (1) identify negative or unrealistic automatic thoughts; (2) evaluate automatic thoughts for accuracy, identify sources of distorted thoughts, recognize the connection between automatic thoughts and emotional/physical shifts; (3) challenge negative, distorted automatic thoughts via "weighing the evidence"; (4) develop new realistic alternative cognitive appraisals; and (5) practice applying new rational appraisals and beliefs.
  Interventions: Behavioral: Cognitive Therapy (CT)
- Mindfulness Meditation (MM) Condition (Active Comparator): Participants randomized to this arm will receive training in mindfulness meditation, specifically Vipassana, which is the form of meditation typically implemented in mindfulness research. With this technique, the emphasis is placed upon developing focused attention on an object of awareness, e.g., the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events.
  Interventions: Behavioral: Mindfulness Meditation (MM)
- Behavioral Activation (BA) Condition (Active Comparator): Participants randomized to this arm will be educated about the role of inactivity and behavioral avoidance in chronic pain and functioning. They will learn how to be aware of the activities they avoid because of pain, and how to set effective goals so that, step by step, they can start being more active and resume some activities they enjoyed in the past but are currently avoiding. Explanation and practice of a set of specific skills - including appropriate pacing skills - to facilitate an increase in appropriate activity level will be provided.
  Interventions: Behavioral: Behavioral Activation (BA)

INTERVENTIONS:
Behavioral: Cognitive Therapy (CT) — The cognitive-restructuring technique will be used to help participants recognize the relationships between thoughts, feelings, behaviors, and pain. This technique will help participants: (1) identify negative or unrealistic automatic thoughts; (2) evaluate automatic thoughts for accuracy, identify sources of distorted thoughts; recognize the connection between automatic thoughts and emotional/physical shifts; (3) challenge negative, distorted automatic thoughts via "weighing the evidence"; (4) develop new realistic alternative cognitive appraisals; and (5) practice applying new rational appraisals and beliefs.
  Arms: Cognitive Therapy (CT) Condition
Behavioral: Mindfulness Meditation (MM) — Participants will receive training in mindfulness meditation, specifically Vipassana, which is the form of meditation typically implemented in mindfulness research. With this technique, the emphasis is placed upon developing focused attention on an object of awareness, e.g., the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events. A standard script will be implemented by the clinician, and participants will be seated in a comfortable yet alert position.
  Arms: Mindfulness Meditation (MM) Condition
Behavioral: Behavioral Activation (BA) — Participants will be educated about the role of inactivity and behavioral avoidance in chronic pain and functioning. They will learn how to be aware of the activities they avoid because of pain, and how to set effective goals so that, step by step, they can start being more active and resume some activities they enjoyed in the past but are currently avoiding. Explanation and practice of a set of specific skills - including appropriate pacing skills - to facilitate an increase in appropriate activity level will be provided.
  Arms: Behavioral Activation (BA) Condition

SUMMARY:
This project will increase our understanding of the mechanisms underlying changes in opioid medication use associated with three psychosocial chronic pain (CP) treatments. These treatments are: (1) Cognitive Therapy (CT), (2) Mindfulness Meditation (MM), and (3) Behavioral Activation (BA). The sample will be adults with CP who are at risk of opioid misuse. The purpose of this study is to understand the specific ways these treatments work for reducing opioid use. In addition, the investigators are interested in examining moderators of treatment response. The findings will potentially inform the future streamlining of psychosocial treatments, as well as the development of algorithms for matching individuals with CP who are at risk for opioid misuse to the specific treatment most likely to efficiently optimize benefit.

DETAILED DESCRIPTION:
This study involves participating in eight videoconference group treatment sessions and telephone interviews over the course of approximately eight to nine months. All study procedures will take place over videoconferencing computer software, online, or by telephone. There are no in-person visits for the study. Participants wear an activity monitor for about two and a half months starting two weeks before treatment begins. They will also complete brief online surveys twice a day, once in the morning and once in the evening, for about two and a half months starting two weeks before treatment begins. These surveys will be completed on a computer, tablet, or smartphone.

Extended Assessments

During the study, participants would also complete four extended assessments with a research staff member. The first interview is completed before treatment begins, the second is completed after treatment ends, the third is completed three months after treatment ends, and the fourth and final is completed six months after treatment ends. The first two extended assessments (Pre- and Post-Treatment) are completed with a research staff member verbally over the telephone. The final two extended assessments (3-month and 6-month Follow-up) may be completed either with a research staff member verbally over the telephone or independently online.

Online Surveys

About two weeks before treatment starts, participants begin doing brief (~2-5 minutes) online surveys twice a day. The online surveys can be completed on a smartphone, tablet, laptop, or desktop computer. Automated notifications in the morning and in the evening remind the participant to complete the brief survey twice a day.

Activity Monitor

Participants wear an activity monitor 24 hours a day for the 2.5-month Monitoring Period (which spans two weeks before treatment to one month after treatment). The activity monitor is worn on the non-dominant wrist, like a wristwatch.

Weekly Interviews

Beginning two weeks prior to treatment, participants will be contacted weekly by a staff member to complete a telephone survey. Participants complete 10 total surveys over the course of 10 weeks, concluding about one month after treatment ends. Each survey takes approximately 10-15 minutes.

Treatment

Participants are randomly assigned to one of the three treatment groups. Treatment consists of eight group treatment sessions completed remotely over a videoconferencing platform. There will be, on average, two sessions per week, and each session will take up to 90 minutes. Each treatment session will take place over the internet on a computer, tablet, or smartphone using the videoconference application. Each session will be led by the same study clinician, who is a trained clinical psychologist. Participants will be required to use a video camera and audio through either a microphone or phone for each group treatment session.

All three treatment interventions will involve educating participants about pain, discussing the impact of pain, and discussing different ways to manage it in hopes of decreasing pain and its impact. The three treatments are: (1) Mindfulness Meditation, (2) Cognitive Therapy, and (3) Behavioral Activation (BA).

Each treatment intervention will have home practice activities to complete between sessions. Home practice activities may include, but are not limited to, creating thought records, listening to pre-recorded guided practices, and keeping track of activities and goals. Participants also receive a treatment workbook with materials to refer to and discuss during the group sessions as well as additional materials to read between sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Meet criteria for having a chronic pain problem (≥3 months, with pain experienced on ≥50% of days in past 6 months);
3. Use of opioid medication in the past week;
4. Daily average opioid analgesic medication use in the past week of ≥20 MMEs;
5. Average intensity of chronic pain ≥3 on a 10-point scale for most days of the previous 3 months;
6. Able to read, speak, and understand English; and
7. Availability of a telephone, webcam, and microphone through computer or telephone, as well as daily internet access.

Exclusion Criteria:

1. Primary pain condition is headache;
2. Severe cognitive impairment;
3. Current alcohol or substance dependence;
4. Active malignancy (e.g., cancer not in remission), terminal illnesses, or serious medical conditions that may interfere with either study participation or with receiving potential treatment benefits (e.g., severe lupus);
5. Inability to walk (defined as unable to walk at least 50 yards), which would limit the ability of participants to benefit from the activation skills intervention;
6. Significant pain from a recent surgery or injury;
7. Pain condition for which surgery has been recommended and is planned;
8. Any planned surgery, procedure, hospitalization, treatment, or event that may conflict with or otherwise influence participation in the study;
9. Currently receiving or had received other psychosocial treatments for any pain condition;
10. Current or past participation in a research study with treatment components that may overlap, conflict, or affect those in the current study;
11. Current or history of diagnosis of primary psychotic or major thought disorder within the past 5 years;
12. Psychiatric hospitalization within the past 6 months;
13. Psychiatric or behavioral conditions in which symptoms were unstable or severe within the past 6 months;
14. Any psychiatric or behavioral issues as noted in the medical record or disclosed/observed during self-report screening that would indicate participant may be inappropriate in a group setting; and
15. Presenting symptoms at the time of screening that would interfere with participation, specifically active suicidal or homicidal ideation with intent to harm oneself or others or active delusional or psychotic thinking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, Ph.D., Principal Investigator — University of Washington; Melissa Day, Ph.D., Principal Investigator — The University of Queensland
Locations (1):
- University of Washington, Ninth and Jefferson Building, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available to interested researchers a data file containing de-identified data used for each published article at the time the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, we will create a data file that includes all variables used in the published article and a list of the variables in the data file (along with variable labels) and mail to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) a CD of the data set (as an SPSS.sav file). Note, though, even though any data files that we share will be stripped of identifiers prior to release for sharing, it remains possible those who access the data could potentially use deduction to identify participants with unusual characteristics or combinations of unusual characteristics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data used for the analyses for any papers published will become available to interested researchers by request after that article is published. Those data will continue to be available for at least five years following the publication of the article.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Day MA, Ciol MA, Ehde DM, Mendoza ME, Borckardt J, Newman AK, Chan JF, Friedly JL, Reed DE 2nd, Drever SA, Burns J, Thorn BE, Jensen MP. The Effects of Psychological Treatments for Chronic Pain on Reducing Opioid Use in People at Risk for Opioid Misuse: A Randomized Feasibility Trial. Pain Pract. 2026 Jan;26(1):e70107. doi: 10.1111/papr.70107. PMID 41230568
- See also: Study website — https://sites.uw.edu/lifestudy/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified primarily via ResearchMatch.org and via coding lists derived from medical records of UW Medicine patients. Other sources of recruitment included social media, the UW Rehabilitation Medicine departmental research participant pool, posted flyers in pain and rehabilitation clinics, clinician referrals, news releases with the UW Newsroom, and a variety of national recruitment strategies.
Pre-assignment Details: N=288 participants were excluded before randomization with 254 not meeting inclusion criteria, 25 unable to be contacted, and 9 declining participation.
Groups:
- Cognitive Therapy (CT) Condition: Participants randomized to this arm will be taught to recognize the relationships between thoughts, feelings, behaviors, and pain. This technique will help participants: (1) identify negative or unrealistic automatic thoughts; (2) evaluate automatic thoughts for accuracy, identify sources of distorted thoughts; recognize the connection between automatic thoughts and emotional/physical shifts; (3) challenge negative, distorted automatic thoughts via "weighing the evidence"; (4) develop new realistic alternative cognitive appraisals; and (5) practice applying new rational appraisals and beliefs.
- Activation Skills (AS) Condition: Participants randomized to this arm will be educated about the role of inactivity and behavioral avoidance in chronic pain and functioning. They will learn how to be aware of the activities they avoid because of pain, and how to set effective goals so that, step by step, they can start being more active and resume some activities they enjoyed in the past but are currently avoiding. Explanation and practice of a set of specific skills - including appropriate pacing skills - to facilitate an increase in appropriate activity level will be provided.
Period: Overall Study
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Activation Skills (AS) Condition
Started | 31 | 29 | 31
Completed | 28 | 26 | 29
Not Completed | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition | Total
Number analyzed (Participants) | 31 | 29 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.4) | 54.4 (11.7) | 51.9 (12.1) | 53.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 25 | 74
  Male | 6 | 5 | 6 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 23 | 24 | 75
  Black/African American | 2 | 4 | 4 | 10
  American Indian/Alaskan Native | 0 | 0 | 1 | 1
  Native Hawaiian/Pacific Islander | 0 | 0 | 1 | 1
  Mixed races | 1 | 2 | 0 | 3
  Unspecified | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 31 | 91
Baseline MME [Mean (Standard Deviation); unit: Morphine milligram equivalent] — Respondents will be asked to provide dosages and frequency of use of any opioid medications taken in the past seven days at baseline. An average daily MME dose taken in the past week will be computed.
  Morphine milligram equivalent | 80.7 (84.7) | 115.8 (215.1) | 75.9 (79.0) | 88.3 (135.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Morphine Milligram Equivalent (MME) Average Daily Dose
Description: Respondents were asked to provide dosages and frequency of use of any opioid medications taken in the past seven days at the time of each telephone assessment. An average daily MME dose taken in the past week was computed for each assessment point, and a categorical variable was calculated to assess change throughout the trial (increase dose, decrease dose, no change).
Time Frame: Collected via phone at pre-treatment (baseline), post-treatment (approximately one month after), and at 3- and 6-months post-treatment (treatment lasted approximately 4 weeks)
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 28 | 26 | 29
participants
  Increase in dose from pre- to post-treatment | 8 | 4 | 5
  Increase in dose from pre- to 3 months post-treatment: number analyzed (Participants) | 26 | 26 | 27
  Increase in dose from pre- to 3 months post-treatment | 5 | 4 | 4
  Increase in dose from pre- to 6 months post-treatment: number analyzed (Participants) | 21 | 23 | 25
  Increase in dose from pre- to 6 months post-treatment | 6 | 7 | 5
  Decrease in dose from pre- to post-treatment | 9 | 14 | 6
  Decrease in dose from pre- to 3 months post-treatment: number analyzed (Participants) | 26 | 26 | 27
  Decrease in dose from pre- to 3 months post-treatment | 12 | 11 | 6
  Decrease in dose from pre- to 6 months post-treatment: number analyzed (Participants) | 21 | 23 | 25
  Decrease in dose from pre- to 6 months post-treatment | 8 | 8 | 6
  No change in dose from pre- to post-treatment | 11 | 8 | 18
  No change in dose from pre- to 3 months post-treatment: number analyzed (Participants) | 26 | 26 | 27
  No change in dose from pre- to 3 months post-treatment | 9 | 11 | 17
  No change in dose from pre- to 6 months post-treatment: number analyzed (Participants) | 21 | 23 | 25
  No change in dose from pre- to 6 months post-treatment | 7 | 8 | 14
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — We hypothesized negligible between condition differences, although within each condition, we hypothesized that each treatment would produce a greater proportion of people decreasing their dose relative to those increasing their dose during treatment; p > .05, Chi-squared

2. Secondary Outcome: Change in Pain Interference (Micro-level)
Description: Change in pain interference with different activities/aspects of life will be measured with five items from the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference item bank. Responses from each item will be summed and converted to a total T-score with a mean of 50 and a standard deviation of 10. Higher scores indicate more self-reported pain interference with different activities/aspects of life. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: Assessed via EMA twice daily during 4-week treatment period, early treatment (1-2 weeks) and late treatment (3-4 weeks) reported
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Early treatment slope | -1.61 (4.78) | -0.13 (5.35) | 0.23 (3.51)
  Late treatment slope | 0.44 (4.54) | 0.81 (7.57) | -1.38 (3.39)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — We hypothesized negligible between condition differences, although within each condition, we hypothesized that each treatment would produce medium effect size improvements; p > .05, ANOVA

3. Secondary Outcome: Change in Affect (Micro-level)
Description: Change in affect will be measured with the Positive and Negative Affect Schedule (PANAS). When assessed with EMA, total scores will range from 1-5 for each affect schedule. A higher positive affect sum score indicates more self-reported positive affect while a lower negative affect sum score indicates less self-reported negative affect. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Positive Affect, early treatment | 0.11 (0.68) | 0.21 (0.64) | -0.01 (0.83)
  Negative Affect, early treatment | -0.15 (0.61) | 0.18 (0.89) | -0.01 (1.01)
  Positive Affect, late treatment | -0.18 (0.66) | 0.15 (0.56) | 0.17 (0.64)
  Negative Affect, late treatment | 0.02 (0.68) | 0.28 (0.66) | -0.04 (0.65)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

4. Secondary Outcome: Change in Physical Function
Description: Change in extent of physical function will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form-4A. Responses are summed and the raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of physical function. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | 0.4 (2.9) | 1.7 (4.1) | 1.5 (6.5)
  Change from pre- to 3 months post-treatment | -0.6 (3.5) | 1.4 (4.7) | 0.9 (3.2)
  Change from pre- to 6 months post-treatment | 0.3 (4.1) | 3.0 (5.2) | 2.3 (4.6)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

5. Secondary Outcome: Change in Sleep Quality
Description: Change in sleep quality will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form-4A. Responses from each item will be summed. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported sleep disturbance. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | -3.9 (8.6) | 0.3 (8.1) | 0.8 (7.8)
  Change from pre- to 3 months post-treatment | -3.4 (6.0) | -0.4 (8.8) | -0.8 (6.8)
  Change from pre- to 6 months post-treatment | -3.3 (6.8) | -0.2 (6.3) | 0.8 (8.5)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

6. Other Pre Specified Outcome: Change in Activity Level (Actigraph, Vector Magnitude Average Counts - Mechanism)
Description: Primary Mechanism Variable
  Change in activity level will be measured by an actigraphy device worn by the participant measuring activity level. In this study, we used the vector magnitude average counts variable, which is the average of all activity counts recorded per minute that the device was worn (i.e., it removes non-wear time from the analysis). Higher activity counts indicate higher intensity activities that day; the minimum possible score theoretically is zero, with no theoretical maximum score. Slopes were calculated by computing the linear regression slopes for the Actigraph collected activity counts.
Time Frame: ActiGraph worn daily during 4-week treatment period, early treatment (baseline-2 weeks) and late treatment (2-4 weeks) reported
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: activity counts
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
activity counts
  Early treatment (at baseline to 2 weeks) | -107353.64 (505760.75) | -20966.51 (437438.18) | 212816.61 (644084.02)
  Late treatment (at 2 weeks to 4 weeks) | 25400.60 (416600.39) | -58278.17 (431604.42) | 93312.68 (607646.06)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

7. Other Pre Specified Outcome: Change in Non-Judgment (Cognitive Process Mechanism, Micro-level)
Description: Primary Mechanism Variable
  Change in non-judgment will be measured with 4 items from the Pain-Related Cognitive Process Questionnaire (PCPQ) Non-Judgmental Scale. Items will be averaged for a mean score from 0-4. Higher mean PCPQ scores indicate higher frequencies of using the adaptive cognitive process of non-judgment in responding to pain. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Early treatment slope | 0.1 (0.6) | 0.1 (0.8) | 0.05 (0.5)
  Late treatment slope | 0.00 (0.5) | 0.00 (0.7) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

8. Other Pre Specified Outcome: Change in Pain Catastrophizing (Cognitive Content Mechanism, Micro-level)
Description: Primary Mechanism Variable
  Change in pain catastrophizing will be measured with items from the University of Washington (UW) Concerns About Pain (CAP) item bank. Responses from the CAP were summed for a total raw score. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of catastrophizing. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Early treatment slope | -2.0 (5.5) | -1.3 (4.4) | -0.8 (4.8)
  Late treatment slope | -0.5 (6.4) | -0.6 (5.5) | -1.1 (4.1)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

9. Other Pre Specified Outcome: Change in Pain Intensity (Mechanism, Micro-level)
Description: Primary Mechanism Variable
  Change in pain intensity of chronic pain will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity. For the EMA data, slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Early treatment slope | -0.1 (1.03) | 0.3 (0.8) | 0.2 (1.1)
  Late treatment slope | 0.2 (1.1) | 0.2 (1.5) | -0.4 (1.1)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

10. Other Pre Specified Outcome: Change in Depression and Anxiety Severity (Mechanism, Macro-level)
Description: Change in depression and anxiety will be measured with the respective Patient-Reported Outcomes Measurement Information System (PROMIS) Short Forms. Responses were summed for a total raw score for depression and anxiety. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of depression and anxiety. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Pre- to post-treatment change in Depression | -3.25 (7.00) | -2.61 (7.83) | -2.55 (6.65)
  Pre- to post-treatment change in Anxiety | -2.23 (7.11) | -2.14 (7.94) | -1.49 (7.21)
  Pre- to 3 months post-treatment change in Depression | -2.41 (6.92) | -2.26 (8.22) | -1.99 (6.45)
  Pre- to 3 months post-treatment change in Anxiety | -1.38 (8.56) | -2.20 (8.97) | -0.45 (8.34)
  Pre- to 6 months post-treatment change in Depression | -2.34 (7.70) | -2.19 (9.38) | -1.87 (7.44)
  Pre- to 6 months post-treatment change in Anxiety | -1.85 (8.42) | -1.41 (9.40) | 0.06 (8.92)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .05, ANOVA

11. Secondary Outcome: Change in Pain Interference (Macro-level)
Description: Change in pain interference with different activities/aspects of life will be measured with five items from the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference item bank. Responses from each item will be summed and converted to a total T-score with a mean of 50 and a standard deviation of 10. Higher scores indicate more self-reported pain interference with different activities/aspects of life. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | -4.8 (7.2) | -6.6 (5.4) | -3.1 (5.9)
  Change from pre- to 3 months post-treatment | -4.6 (5.7) | -2.9 (5.2) | -2.1 (5.9)
  Change from pre- to 6 months post-treatment | -4.0 (6.1) | -3.0 (6.2) | -1.7 (5.9)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

12. Secondary Outcome: Change in Affect (Macro-level)
Description: Change in affect will be measured with the Positive and Negative Affect Schedule (PANAS). When assessed via phone, responses from the positive affect items will be summed for a total positive score ranging from 5-25 while responses from the negative affect items will be separately summed for a total negative score ranging from 5-25. When assessed with EMA, total scores will range from 1-5 for each affect schedule. A higher positive affect sum score indicates more self-reported positive affect while a lower negative affect sum score indicates less self-reported negative affect. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Positive Affect, change from pre- to post-treatment | 0.6 (3.3) | 1.8 (3.0) | 0.4 (2.3)
  Negative Affect, change from pre- to post-treatment | -2.1 (3.8) | -1.5 (4.4) | -0.6 (2.6)
  Positive Affect, change from pre- to 3 months post-treatment | -0.3 (3.4) | 1.0 (3.7) | -1.2 (3.5)
  Negative Affect, change from pre- to 3 months post-treatment | -1.8 (3.3) | -1.0 (4.2) | 0.5 (3.2)
  Positive Affect, change from pre- to 6 months post-treatment | 0.3 (3.4) | 0.7 (3.2) | -0.9 (3.3)
  Negative Affect, change from pre- to 6 months post-treatment | -1.8 (4.2) | 0.3 (3.8) | 0.4 (4.6)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

13. Other Pre Specified Outcome: Change in Activity Level (Self-report Mechanism, EMA)
Description: Secondary Mechanism Variable
  Self-reported change in activity level will be measured via the Godin Leisure-Time Exercise Questionnaire (GLTEQ). The daily EMA items asked how many times that day did the participant engage in >15mins of strenuous exercise, >15mins of moderate exercise and >15mins of mild exercise. The total frequencies for each category for a week were summed, and this scoring formula was applied to calculate overall units of activity: Activity Score = (9 x Freq. of Strenuous)+(5 x Freq. of Moderate)+(3 x Freq. of Mild). The lowest possible score is zero, while no theoretical maximum score exists. Higher scores indicate higher levels of activity. Slopes (reported unit of measure) were calculated by computing the linear regression slopes, which are equivalent in meaning and magnitude to change scores.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
scores on a scale
  Early treatment slope | 3.3 (25.4) | -1.0 (23.2) | -0.3 (20.5)
  Late treatment slope | -2.1 (16.5) | 6.6 (19.8) | 8.0 (21.2)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

14. Other Pre Specified Outcome: Change in Activity Level (Self-report Mechanism, Telephone Assessed)
Description: Secondary Mechanism Variable
  Self-reported change in activity level will be measured via the Godin Leisure-Time Exercise Questionnaire (GLTEQ). Participants were asked how many times in the past 7-days did they engage in >15mins of strenuous exercise, >15mins of moderate exercise and >15mins of mild exercise. This scoring formula was applied to calculate overall units of activity: Activity Score = (9 x Freq. of Strenuous)+(5 x Freq. of Moderate)+(3 x Freq. of Mild). The lowest possible score is zero, while no theoretical maximum score exists. Higher scores indicate higher levels of activity. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | 13.31 (41.67) | 11.63 (45.34) | 20.65 (51.77)
  Change from pre- to 3 months post-treatment | 16.40 (151.63) | 1.83 (53.54) | 45.75 (193.01)
  Change from pre- to 6 months post-treatment | 0.89 (114.42) | 0.59 (34.73) | 0.05 (33.12)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

15. Other Pre Specified Outcome: Change in Non-Judgment (Cognitive Process Mechanism, Macro-level)
Description: Primary Mechanism Variable
  Change in non-judgment will be measured with items from the Pain-Related Cognitive Process Questionnaire (PCPQ) Non-Judgmental Scale. The full 6-item scale will be used. Items will be averaged for a mean score from 0-4. Higher mean PCPQ scores indicate higher frequencies of using the adaptive cognitive process of non-judgment in responding to pain. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | 0.43 (1.14) | 0.45 (1.19) | 0.48 (1.18)
  Change from pre- to 3 months post-treatment | 0.39 (1.01) | 0.35 (1.34) | 0.57 (1.04)
  Change from pre- to 6 months post-treatment | 0.36 (0.98) | 0.41 (1.24) | 0.46 (1.20)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

16. Other Pre Specified Outcome: Change in Pain Catastrophizing (Cognitive Content Mechanism, Macro-level)
Description: Primary Mechanism Variable
  Change in pain catastrophizing will be measured with items from the University of Washington (UW) Concerns About Pain (CAP) item bank. Responses from the CAP were summed for a total raw score. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher levels of catastrophizing. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Change from pre- to post-treatment | -7.12 (8.45) | -6.91 (9.85) | -8.28 (8.12)
  Change from pre- to 3 months post-treatment | -6.72 (9.32) | -4.70 (8.76) | -7.97 (9.49)
  Change from pre- to 6 months post-treatment | -5.47 (10.29) | -5.82 (9.59) | -6.56 (9.62)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

17. Other Pre Specified Outcome: Change in Pain Intensity (Mechanism, Macro-level)
Description: Primary Mechanism Variable
  Change in pain intensity of chronic pain will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity. Change scores were then calculated for the pre- and post-treatment and 3-month and 6-month follow-up data.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
Number analyzed (Participants) | 31 | 29 | 31
change score on a scale
  Pre- to post-treatment change | -0.99 (1.80) | -1.18 (2.13) | -1.29 (1.90)
  Pre- to 3 months post-treatment change | -0.90 (1.70) | -0.82 (1.89) | -1.40 (2.23)
  Pre- to 6 months post-treatment change | -0.96 (1.87) | -1.03 (1.99) | -1.09 (2.03)
Statistical Analysis 1: Comparison: Cognitive Therapy (CT) Condition vs Mindfulness Meditation (MM) Condition vs Behavioral Activation (BA) Condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p > .05, ANOVA

ADVERSE EVENTS:
Time Frame: All participants were monitored/assessed for adverse events from enrollment through study completion, which was an average of 9 months.
Description: Adverse events (AEs) were self-reported by participants and documented in an electronic regulatory event. The majority of AEs reported by participants were conveyed to researchers without prompt. AE monitoring occurred at the beginning of each treatment session with therapists asking if anyone had any negative effects attributed to the treatment. Any concerns that met the definition of an AE were documented. AEs were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Cognitive Therapy (CT) Condition | Mindfulness Meditation (MM) Condition | Behavioral Activation (BA) Condition
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 1/31
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/29 | 4/31
Other Adverse Events (participants affected / at risk) | 15/31 | 15/29 | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Therapy (CT) Condition (N=31) | Mindfulness Meditation (MM) Condition (N=29) | Behavioral Activation (BA) Condition (N=31)
Hospitalization related to new infection/illness (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) — Not study related
Hospitalization due to new/existing respiratory illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Not study related
Hospitalization due to new/existing immune system illness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
Hospitalization related to a surgery/procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Not study related
Hospitalization related to suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Hospitalization due to illness of multiple organ systems (General disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Therapy (CT) Condition (N=31) | Mindfulness Meditation (MM) Condition (N=29) | Behavioral Activation (BA) Condition (N=31)
Increase in existing chronic pain symptoms related to a study procedure (Social circumstances) | 1 (1) | 1 (1) | 2 (2)
Increase in pain due to new injury/accident (Injury, poisoning and procedural complications) | 4 (6) | 4 (4) | 5 (6) — Not study related
New/worsening symptoms related to medical procedure/treatment (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not study related
New/worsening skin irritation/rash related to wearing study ActiGraph device (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 4 (4)
New/worsening respiratory symptoms/illness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 3 (3) — Not study related
New/worsening symptoms related to the endocrine system (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — Not study related
New/worsening psychological discomfort related to a study procedure (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
New/worsening gastrointestinal symptoms/illness (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) — Not study related
Increase in existing chronic pain symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 3 (3) — Not study related
New/worsening sleep problem (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Not study related
New/worsening headache/migraine (Nervous system disorders) | 1 (1) | 4 (5) | 2 (2) — Not study related
New/worsening symptoms related to multiple organ systems (General disorders) | 1 (1) | 0 (0) | 1 (1) — Not study related
New surgery/medical procedure (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) — Not study related
New/worsening infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Not study related
New neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Not study related
New/worsening urinary illness/infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
New/worsening kidney related symptoms/illness (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) — Not study related
New/worsening neurological symptoms/illness (not migraine) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Victim of assault (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Not study related
Adverse reaction related to treatment/medication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Not study related
New/worsening cardiovascular symptoms/illness (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
New/worsening psychological distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) — Not study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03916276/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03916276/SAP_001.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03916276/ICF_002.pdf